CLINICAL TRIAL: NCT03965585
Title: Office Hysteroscopy in the Infertility Work-out: the Role of Endometrial Hyperplasia in Southern Italian Women
Brief Title: Office Hysteroscopy in Infertility Work-out: the Role of Endometrial Hyperplasia in Southern Italian Women
Status: Completed | Type: Observational
Sponsor: University of Campania Luigi Vanvitelli (Other)
Responsible Party: Principal Investigator, Prof. Pasquale De Franciscis, Associate Professor, University of Campania Luigi Vanvitelli
Other Study IDs: N.593
Record Dates: First submitted 2019-05-21; First posted 2019-05-29 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Infertility, Female; Endometrial Hyperplasia; PCOS
MeSH Terms: conditions — Infertility, Female; Endometrial Hyperplasia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Primary Infertility: Women with a diagnosed primary infertility undergoing hysteroscopy before IVF.
  Interventions: Procedure: in-office hysteroscopy
- Secondary Infertility: Women with a diagnosed secondary infertility undergoing hysteroscopy before IVF.
  Interventions: Procedure: in-office hysteroscopy
- Recurrent miscarriages: Women with recurrent miscarriages undergoing hysteroscopy before IVF.
  Interventions: Procedure: in-office hysteroscopy

INTERVENTIONS:
Procedure: in-office hysteroscopy — in-office hysteroscopy with miniaturized instruments

SUMMARY:
To assess the prevalence of endometrial hyperplasia (EH), endometrial intraepithelial neoplasia (EIN) and endometrial carcinoma between obese and not obese women undergoing IVF techniques for primary or secondary infertility.

DETAILED DESCRIPTION:
Endometrial cancer and pre-neoplastic diseases represent the most incident gynecologic malignant pathologies found in women.1 Although diagnosed in postmenopausal patients, it can be also found in younger patients, especially when associated with some risk factors. Those include weight gain and lifestyle habits, such as consumption of fatty foods that increase estrogen levels. The positive association be- tween infertility and EC is well established. Infertile women with irregular menstrual periods, oligomenorrhea, or chronic anovulation have a risk of developing

A prospective cohort study conducted at "Fertility Center, OB/GYN Unit, Department of Woman, Child and General and Specialized Surgery, University of Campania "Luigi Vanvitelli", Naples, Italy".

ELIGIBILITY:
Inclusion Criteria:

* Women undergoing office hysteroscopy prior to IVF techniques

Exclusion Criteria:

* Severe comorbidities (i.e. cardiac, metabolic, neurologic diseases)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Southern Italian women eager for children who are set for infertility work-up at a tertiary university hospital
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2019-01-02 (Actual); Primary Completion 2019-04-21 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
Prevalence of endometrial hyperplasia | 12 months
Hormonal levels | 12 months

SECONDARY OUTCOMES:
Operator's learning curve with cumulative summation test (questionnaire) | 12 months
  assess the learning curve (LC) using cumulative summation test for learning curve (LC-CUSUM).

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Woman, Child and General and Specialized Surgery, University of Campania "Luigi Vanvitelli", Naples, Italy

IPD SHARING:
Plan to Share IPD: No